CLINICAL TRIAL: NCT00187538
Title: Effect of Dietary Protein Source on Calcium Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H9291-19207-05
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Calcium Metabolism
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Behavioral: Dietary
- 2 (Active Comparator)
  Interventions: Behavioral: Dietary
- 3 (Active Comparator)
  Interventions: Behavioral: Dietary
- 4 (Active Comparator)
  Interventions: Behavioral: Dietary

INTERVENTIONS:
Behavioral: Dietary — dietary

SUMMARY:
Osteoporosis is a major health concern worldwide. While there are drugs available for the treatment and prevention of osteoporosis, they are not practical for population-wide prevention efforts. Demonstrating the effectiveness of safe and widely available dietary interventions to prevent osteoporosis could have important public health ramifications. Different food sources of dietary protein may have different effects on bone metabolism. Animal foods provide a dietary acid load that may lead to negative calcium balance and increased bone resorption. In contrast, vegetable sources of protein, while providing some acid due to their protein content, provide proportionally more base that counters the dietary acid load. The effect of dairy products, which are rich in animal protein but also contain potential base precursors not found in vegetable foods, has not been established. Finally, soy protein sources may have a dual benefit: soy foods provide base precursors as well as plant estrogens that may have a beneficial effect on bone. We are resubmitting this proposal to randomize postmenopausal women to one of four diets equal in calories, protein, calcium, and sodium. The diets will differ by having 80 percent of the protein from one of four sources: non-dairy animal, vegetable, dairy, or soy foods, resulting in significant differences among the diets in acid, base, and isoflavone content. All food will be prepared and provided by the General Clinical Research Center. The subjects will consume the diets for 6 weeks with measurements of acid-base status, isoflavone excretion, and calcium metabolism. This will be the first intervention study to examine the effect of different sources of dietary protein in whole foods on calcium metabolism. Eventually our findings could have substantial public health implications and provide a widely available and low risk means to help prevent osteoporosis.

DETAILED DESCRIPTION:
Demonstrating the effectiveness of safe and widely available dietary interventions to prevent osteoporosis could have important public health ramifications. Different food sources of dietary protein may have different effects on bone metabolism. Animal foods provide a dietary acid load that may lead to negative calcium balance and increased bone resorption. In contrast, vegetable sources of protein, while providing some acid due to their protein content, provide proportionally more base that counters the dietary acid load. The effect of dairy products, which are rich in animal protein but also contain potential base precursors not found in vegetable foods, has not been established. Finally, soy protein sources may have a dual benefit: soy foods provide base precursors as well as plant estrogens that may have a beneficial effect on bone. We are resubmitting this proposal to randomize postmenopausal women to one of four diets equal in calories, protein, calcium, and sodium. The diets will differ by having 80 percent of the protein from one of four sources: non-dairy animal, vegetable, dairy, or soy foods, resulting in significant differences among the diets in acid, base, and isoflavone content. All food will be prepared and provided by the General Clinical Research Center. The subjects will consume the diets for 6 weeks with measurements of acid-base status, isoflavone excretion, and calcium metabolism. This will be the first intervention study to examine the effect of different sources of dietary protein in whole foods on calcium metabolism. Eventually our findings could have substantial public health implications and provide a widely available and low risk means to help prevent osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

Healthy postmenopausal women

Exclusion Criteria:

No meds affecting bone Normal renal, GI, hepatic function

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2002-02; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
calcium metabolism | after 8 weeks of diet

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Sellmeyer, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Gonciulea AR, Sellmeyer DE. The effect of dietary protein source on serum lipids: Secondary data analysis from a randomized clinical trial. J Clin Lipidol. 2017 Jan-Feb;11(1):46-54. doi: 10.1016/j.jacl.2016.09.014. Epub 2016 Oct 3. PMID 28391910